CLINICAL TRIAL: NCT03010761
Title: Establishment of Cessation Therapy by Clinical Trials for Subjects With Betel-quid Dependence and Oral Pre-cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: all participants finished the trial
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C103RE1059
Record Dates: First submitted 2016-07-25; First posted 2017-01-05 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Addiction
Keywords: addiction; betel-quid; drug therapy; clinical trial
MeSH Terms: conditions — Behavior, Addictive | interventions — Escitalopram; Moclobemide; bisaramil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- medication pills 1: escitalopram 10mg (Experimental): 10mg once daily, 8 weeks
  Interventions: Drug: escitalopram
- medication pills 2: moclobemide 150mg (Experimental): 150mg once daily, 8 weeks
  Interventions: Drug: Moclobemide
- medication pills 3: Placebo - Cap (Experimental): placebo once daily, 8 weeks
  Interventions: Drug: Placebo - Cap

INTERVENTIONS:
Drug: escitalopram — antidepressant use for the betel-quid abstinence
  Other Names: Lexapro
  Arms: medication pills 1: escitalopram 10mg
Drug: Moclobemide — antidepressant use for the betel-quid abstinence
  Other Names: yutac
  Arms: medication pills 2: moclobemide 150mg
Drug: Placebo - Cap — Placebo - Cap
  Arms: medication pills 3: Placebo - Cap

SUMMARY:
No medication existed for BQ dependence. No clinical trials existed for the drug therapy. Previous study showed that BQ possessed the antidepressant effect via pathway of monoamine oxidase A (MAO-A). An animal model also found that the arecoline from BQ has a property as MAO-A inhibitor. Therefore, the investigators hypothesized that inhibition of the MAO-A or antidepressants might reduce the BQ addiction severity.

The investigators will conduct the randomization and double blinded with placebo controlled study with 90 participants with BQ dependence from the Family Medicine and ear, nose, and throat (ENT) outpatient department (OPD). All participants shall agree the informed consent. The range of age is from 18 to 65 years old. The participants are diagnosed as BQ use disorder without other psychiatry co-morbidity, according to the Diagnostic and Statistical Manual (DSM)-V criteria. Those who have severe physical illness, psychiatric illness, and other substance use disorder except cigarettes are excluded. All participants receive the semi-structure interview by DSM-V, International Classification of Diseases (ICD)-10, and Mini International Neuropsychiatric Interview by the psychiatrist. Before the intervention, the participants will finish their basic data, daily amount of cigarettes, betel nut, medical history and psycho-social rating scales. Next, in addition to counseling, the investigators will continue or modify the optimal antidepressants based on the previous results.

The investigators will evaluate their BQ use condition as what has been measured in the natural observation study of the first year. The investigators will check the outcome measurement by visual analog scale, betel quid withdrawal severity scale, Yale-Brown Obsessive-Compulsive (Y-BOCS) - betel quid (BQ) scale. The investigators also followed their hamilton depression scale; Beck depression index; and Beck anxiety index in the baseline, 2nd, 4th, 6th , and 8th week. The investigators also obtained the participants' gene type if the participants also agree for the prediction of oral cancers.

DETAILED DESCRIPTION:
We'll conduct the betel-quid (BQ) dependence clinical trial since 2016. Eligible cases will be enrolled for the following 8 week double-blinded placebo controlled trial. The groups will be divided into three groups. Outcome measures include BQ use condition, addiction severity rating scale, emotional rating scale including Beck Anxiety Index (BAI), Beck Depression Index (BDI), Hamilton Depression Scales (HAMDs), and urine BQ metabolites.

ELIGIBILITY:
Inclusion Criteria:

* DSM-V criteria suitable for betelnut use disorder
* No severe physical disorder
* No major psychiatric illness
* Chinese Speaker

Exclusion Criteria:

* Severe physical disorder
* Major psychiatric illness
* Inability to understand the whole protocol

Ages: 14 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
betelnut use severity rating scale for addiction severity of betelnut | 8 weeks
  The betelnut severity rating scale is a questionnaire rated by the psychiatrist or trained psychologist/nurse, containing 21 yes or no questions about betelnut use

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale for depression | 8 weeks
  for depression
Beck depression index, copyrighted in Chinese (The Psychological Cooperation, Harcourt Brace& Company) | 8 weeks
  self-rating for depression
Beck anxiety index, copyrighted in Chinese (The Psychological Cooperation, Harcourt Brace& Company) | 8 weeks
  self-rating for anxiety
betelnut use Yale-Brown Obsessive Compulsive Disorder-like Scale for the craving status | 8 weeks
  Yale-Brown Obsessive Compulsive Disorder-like Scale, translated in Chinese and betelnut use craving form, a questionnaires containing 10 questions rated by the psychiatrist or trained psychologist/nurse, severity from 0-4
betelnut metabolites urinary analysis | 8 weeks
  arecoline, arecaidine, and N-methylnipecotic acid checked by liquid chromatography mass spectrometry (LC-MS)

CONTACTS AND LOCATIONS:
Overall Officials: Ko Ying-Chin, PHD, Study Director — China Medical University Hospital

IPD SHARING:
Plan to Share IPD: Yes